CLINICAL TRIAL: NCT04945057
Title: AKTIBIPO-VALIDATION: A Study to Validate Benefits of Mindpax System in Managing Bipolar Disorder
Acronym: VAL1M
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Collaborators: Mindpax s.r.o., Czech Republic (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AKTIBIPO-VALIDATION
Record Dates: First submitted 2021-06-01; First posted 2021-06-30 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Participants previously followed in the AKTIBIPO study and newly admitted participants (DeNovo) are included. Participants are followed over 12 months in the programme, collecting primary outcome every 3 months. Some long-term secondary outcomes are compared to values from the equivalent amount of time in the preceding AKTIBIPO study. The newly admitted DeNovo participants are followed for additional 3 months prior to starting the digital programme to collect outcome data from a non-interventional comparison period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): All participants will use the Mindpax mobile application, wear the wrist accelerometer and fill in weekly self-assessments. All participants will obtain weekly health tips (general psychoeducation) and additional individualized targeted tips when the system detects deviation from individual mood, activity and sleep patterns.
  Participants, who did not participate in the previous AKTIBIPO study (DeNovo) will complete additional 3 months of actigraphy and self-evaluation monitoring with research version of the Mindpax application, providing limited feedback and no health tips.
  Interventions: Device: Mindpax monitoring system

INTERVENTIONS:
Device: Mindpax monitoring system — All participants will use the Mindpax mobile application, wear the wrist accelerometer and fill in weekly self-assessments. All participants will obtain weekly health tips (general psychoeducation) and additional individualized targeted tips when the system detects deviation from individual mood, activity and sleep patterns, during the active 12 months of followup.

SUMMARY:
The aim of the AKTIBIPO VALIDATION study is to evaluate the effect of the Mindpax monitoring and microeducation system in patients with bipolar disorder (BD). Up to 130 participants (BD patients) who participated previously in the observational AKTIBIPO study, as well as new patients (DeNovo) will be enrolled for a follow-up period of 12 months. All participants will wear the wrist actigraphy device and use the Mindpax mobile application on their mobile phone. Through the application, the patients will fill in the weekly mood self assessment questionnaire (ASERT) and receive evidence-based health microeducations aimed at understanding the bipolar disorder and associated risk factors. Apart from general psychoeducation, the participants will receive additional individualized targeted health microeducation when the system detects deviation from individual patterns of mood, activity and sleep. The outcomes will evaluate the subjective and objective impact of system usage on self-reported and clinical outcomes.

DETAILED DESCRIPTION:
Study procedure

Up to 130 participants (BD patients) who participated previously in the observational AKTIBIPO study and patients with no history of using the Mindpax system (DeNovo) will be enrolled for a follow-up period of 12 months (+ 3 additional months for DeNovo patients). All participants will wear the wrist actigraphy device (Mindpax) at all times and use the Mindpax mobile application. At enrollment and study completion, the participants will sign the informed consent and undergo evaluation using the MADRS (Montgomery-Asberg depression rating scale) and YMRS (Young mania rating scale) scales.

Collected data

At baseline, i.e. at enrollment to the digital programme (M0) and every three months (M3,M6,M9,M12), the participants will fill in a series of self-assessment questionnaires: the Q-les-Q (the Quality of life Enjoyment and Satisfaction Questionnaire), HLS-CZ-12 (Health literacy survey), WHODAS 2.0 CZ (the WHO disability assessment schedule), BMQ-CZ (Beliefs about medicines questionnaire) and MARS-CZ (the Medication adherence report scale). The patients will also be evaluated using the CGI-S (Clinical global impression, M0-M12). The psychosocial and clinical events (hospitalizations, relapses), current medication and illness history will be collected throughout the study (M0-M12).

The DeNovo patients with no history of using the Mindpax application will complete additional 3 months of actigraphy and self-assessment monitoring with no intervention and limited feedback (mirror period), prior to visit M0. At entering this observational period, the same set of aforementioned instruments will be collected (visit M-3).

Study endpoints

The primary endpoint is the change in Q-les-Q score at M12, compared to M0. Secondary endpoints include: i) higher health status (lower number of hospitalization days, compared to the same amount of time in the preceding AKTIBIPO study or mirror period for DeNovo patients), ii) lower subjectively rated symptom level (compared to the same amount of time in the preceding AKTIBIPO study or mirror period), iii) higher rate of health literacy at M12, compared to M0, and iv) Higher treatment adherence and better understanding to medication at M12, compared to M0.

Microeducation

* During the study, microeducation messages will be delivered to patients via Mindpax smartphone app on a regular basis (at least once a week, maximum two messages per week).
* This approach will aim at well-being, coping with stress, increasing the regularity and stabilization of social rhythms, daily routines and therapy adherence. The main focus is to enhance role functioning in the society and workspace, and decrease the likelihood of another mood episodes among patients in a symptomatic illness stage.
* Generic microeducational messages will address a wide array of stress-coping and interpersonal problem areas such as grief for "losing" the healthy self and disagreements with others, promoting the importance of therapy adherence, addressing transitions that can affect the patient's normal routine, supplying information on managing the bipolar illness, and providing tools for relapse prevention
* Two types of alert scores will be calculated for duration of sleep and overall activity. Based on this alerting system, target microeducative messages will be consequently generated and delivered on the participant's smartphone to help patients change their maladaptive behavior by reducing current sleep/wake and daily activity irregularity and avoid behaviors that may adversely affect social rhythms.
* In a meantime, digital diary smartphone feedback will provide continuously upgraded infographics on variability of daily activities such as wake time, bed time, sleep onset, sleep regularity and inter-daily variability in those parameters.
* This circadian feedback feature will inform patients to what extent the past microeducative messages influenced their daily routines. This way, a feedback information will encourage participants to change their behavior by showing the impact that corrective behavior had on their mood. App feedback and microeducative content could help prevent recurrences by helping the subject to recognize and modify their future behaviors

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a diagnosis of bipolar disorder (BD, F31.x)
* between 18 to 65 years old.
* Participants with acceptable compliance in the past AKTIBIPO400 study: completeness of activity data and weekly mood reporting data at least 50% each.
* Newly admitted patients (DeNovo): currently treated for BD, ability to provide psychiatric hospitalization history provided from medical health record or health insurance records.

Exclusion Criteria:

* Organic mental disorder
* mental disorder due to psychoactive substance use,
* current hospitalization or mood episode at admission, measured by the Montgomery-Åsberg Depression rating scale (MADRS) ≥ 19 or Young Mania Rating Scale (YMRS) ≥ 19 at admission.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life (Q-LES-Q) at 12 months | 12 months
  Change from baseline in the Quality of Life Enjoyment and Satisfaction Questionnaire at final visit 12 months from enrolment.

SECONDARY OUTCOMES:
Change in quality of life (Q-LES-Q) at 6 months | 6 months
  Change from baseline in the Quality of Life Enjoyment and Satisfaction Questionnaire 6 months from enrolment.
Change in level of disability (WHODAS) at 12 months | 12 months
  Change from baseline in the WHO Disability Assesment Schedule 2.0 at final visit 12 months from enrolment.
Change in level of disability (WHODAS) at 6 months | 6 months
  Change from baseline in the WHO Disability Assesment Schedule 2.0 at 6 months from enrolment.
Lower number of hospitalization days during 12 months o of followup, compared to a preceding study | up to 12 months, mirror design
  The number of hospitalization days during the 12 months follow-up in the study as reported by the patient/caring psychiatrist, compared to the mirror period.
  The mirror period is defined as the last time window of the preceding AKTIBIPO study which fulfilled the data completeness criteria (i.e. at least 50% valid actigraphy days and at least 50% completed weekly ASERT questionnaires) and has equal length to the followup in the AKTIBIPO-VALIDATION study. If the participant exists the study prematurely, the last period of equal length of the AKTIBIPO study, fulfilling the criteria, will be used.
Lower number of hospitalization days during first 6 months of followup, compared to a preceding study | 6 months, mirror design
  The number of hospitalization days during the first 6 months follow-up in the study as reported by the patient/caring psychiatrist, compared to the mirror period.
  The mirror period is defined as the last time window of the preceding AKTIBIPO study which fulfilled the data completeness criteria (i.e. at least 50% valid actigraphy days and at least 50% completed weekly ASERT questionnaires) and has equal length to the followup in the AKTIBIPO-VALIDATION study. If the participant exists the study prematurely, the last period of equal length of the AKTIBIPO study, fulfilling the criteria, will be used.
Lower mean value of the subjectively rated symptom level using the Aktibipo SElf-RaTing (ASERT) questionnaire at 12 months | up to 12 months, mirror design
  Difference of the mean value of the total score of the subjectively rated symptom level using the Aktibipo SElf-RaTing (ASERT) questionnaire (Anýž. J., 2021) during the 12 months of followup compared to the mirror period
  The mirror period is defined as the last time window of the preceding AKTIBIPO study which fulfilled the data completeness criteria (i.e. at least 50% valid actigraphy days and at least 50% completed weekly ASERT questionnaires) and has equal length to the followup in the AKTIBIPO-VALIDATION study. If the participant exists the study prematurely, the last period of equal length of the AKTIBIPO study, fulfilling the criteria, will be used.
Lower mean value of the subjectively rated symptom level using the Aktibipo SElf-RaTing (ASERT) questionnaire at 6 months | 6 months, mirror design
  Difference of the mean value of the total score of the subjectively rated symptom level using the Aktibipo SElf-RaTing (ASERT) questionnaire (Anýž. J., 2021) during the first 6 months of followup compared to the mirror period
  The mirror period is defined as the last time window of the preceding AKTIBIPO study which fulfilled the data completeness criteria (i.e. at least 50% valid actigraphy days and at least 50% completed weekly ASERT questionnaires) and has equal length to the followup in the AKTIBIPO-VALIDATION study. If the participant exists the study prematurely, the last period of equal length of the AKTIBIPO study, fulfilling the criteria, will be used.
Higher rate of health literacy (HLS-12-CZ) at 12 months | 12 months
  Higher value of the as measured by the Health literacy survey HLS-12-CZ questionnaire at 12 months, compared to baseline.
Higher rate of health literacy (HLS-12-CZ) at 6 months | 6 months
  Higher value of the as measured by the Health literacy survey HLS-12-CZ questionnaire at 6 months, compared to baseline.
Higher value of medication adherence report scale (MARS) at 12 months | 12 months
  The difference in the total score of the Medication Adherence Report Scale (MARS) at 12 months of followup, compared to baseline
Higher value of medication adherence report scale (MARS) at 6 months | 6 months
  The difference in the total score of the Medication Adherence Report Scale (MARS) at 12 months of followup, compared to baseline
Higher rate of beliefs about medicines questionnaire (BMQ) at 12 months | 12 months
  The difference of the total score of the Beliefs about medicines questionnaire (BMQ-CZ) at 12 months, compared to baseline.
Higher score of beliefs about medicines questionnaire (BMQ) at 6 months | 6 months
  The difference of the total score of the Beliefs about medicines questionnaire (BMQ-CZ) at 6 months, compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health, Klecany, Czechia

IPD SHARING:
Plan to Share IPD: No